CLINICAL TRIAL: NCT05869916
Title: The Effect of Psychological First Aid Intervention on Stress and Resilience in Volunteers Working in Kahramanmaraş Centered Earthquakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Esra Bekircan, lecturer, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Psychological First Aid
Record Dates: First submitted 2023-05-01; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Psychological Resilience; Stress; Earthquake
Keywords: post traumatic stress disorder; psychological first aid; psychological resilience; earthquake victims
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psychological First Aid

STUDY DESIGN:
Intervention Model Description: This research is a single-blind randomized controlled experimental study to determine the effect of online psychological first aid intervention on the stress and resilience levels of volunteers who took part in the earthquake.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Volunteers working in the provinces affected by the earthquake were reached by snowball sampling (Patton, 1990). In order to provide blinding, only one of the researchers interviewed individuals by snowball sampling method. 34 people who wanted to be included in the study and were included in the inclusion criteria were assigned to the experimental and control groups by a simple random sampling method by a statistician who was not included in the study. In order to prevent contamination and bias between the groups and the researcher who applied the psychological first aid, attention was paid to avoid any interaction before the application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In this study, the "Psychological First Aid: A Guide for Field Workers" program published by the World Health Organization in 2011 was adapted to the needs and culture of the region/people where the research will be conducted. Psychological First Aid training was given by the psychiatric nurse participating in the study after a two-day training organized by the Psychiatric Nursing Association.
  Interventions: Behavioral: psychological first aid
- control group (No Intervention): No interference

INTERVENTIONS:
Behavioral: psychological first aid — The effect of psychological first aid on earthquake victims was measured using the resilience scale and the secondary traumatic stress scale.
  Arms: experimental group

SUMMARY:
Purpose: It was aimed to compare the effectiveness of online psychological first aid intervention on stress and psychological resilience in volunteers who took part in earthquakes.

Method: This is a single-blind randomized controlled experimental study conducted to determine the effect of online psychological first aid intervention on the stress and resilience levels of volunteers who took part in the earthquake.

DETAILED DESCRIPTION:
In this study, it is aimed to compare the effectiveness of the online psychological first aid intervention on stress and psychological resilience given to the volunteers working in various provinces (11 provinces) affected by the Kahramanmaraş Centered Earthquakes.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering in the earthquake zone,
* Not having a perception disorder that will prevent communication,
* To volunteer to participate in the research.

Exclusion Criteria:

* Having a communication barrier,
* Not wanting to be involved in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
1st hypothesis | 2 weeks
  The resilience level of the experimental group who received psychological first aid intervention was increased by using the psychological resilience scale.
2nd hypothesis | 2 weeks
  The stress level of the experimental group, which received psychological first aid intervention, was reduced by using the secondary stress scale psychological.

CONTACTS AND LOCATIONS:
Overall Officials: galip usta, 2, Study Director — galipusta@trabzon.edu.tr; kemal torpuş, 3, Study Director — kemaltorpus@artvin.edu.tr
Locations (1):
- The data of the study were collected between February 20, 2023 and March 20, 2023 in the form of group interviews by applying online psychological first aid to volunteers working in Kahramanmaraş Centered Earthquakes that occurred in Turkey on Monday, Feb, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Model of the Research This research is a single-blind randomized controlled experimental study to determine the effect of online psychological first aid intervention on the stress and resilience levels of volunteers who took part in the earthquake. In this model, there is an experimental group formed by randomization and a control group.